CLINICAL TRIAL: NCT04923152
Title: Effects of High- or Moderate-Dose Statin on 1-Year Major Adverse Cardiovascular Events (MACE) Post Percutaneous Coronary Interventions
Brief Title: Effective Dose of Statin Post PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, Professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SUMS.MED.REC.1398.620
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Statin Dose
Keywords: PCI; Stable Angina; statin therapy
MeSH Terms: conditions — Angina, Stable | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: double blind randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group A, group B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate dose statin (Experimental): Patients 1 month post PCI, allocated to 5 mg rosuvastatin per day
  Interventions: Drug: moderate statin dose
- high dose statin (Active Comparator): patients 1 month post PCI, allocated to 40 mg rosuvastatin
  Interventions: Drug: high dose statin

INTERVENTIONS:
Drug: moderate statin dose — 5 mg rosuvastatin per day
  Arms: moderate dose statin
Drug: high dose statin — 40 mg rosuvastatin per day
  Arms: high dose statin

SUMMARY:
In this study post coronary stenting patients, were enrolled to receive moderate dose versus high dose statin for 1 year, and the result of major adverse cardiovascular events were recorded

DETAILED DESCRIPTION:
In this randomized double-blind clinical trial, the study population was all patients with a recent history of PCI who referred to the professor kojuri cardiovascular clinic for the first post-procedure visit. In the first visit, patients were randomly divided into two groups Both groups were treated with Rosuvastatin 40 mg as high potency statin for one month after PCI. In the first group, after one month, the statin level changed to Rosuvastatin 5 mg daily (moderate intensity). In the second group, 40 mg of Rosuvastatin was continued for one year. Then, the participants were evaluated in terms of MACEs, including any hospitalization due to acute coronary syndrome, as well as history of stroke and myocardial Infarction, subsequent unplanned revascularization and cardiac death. The HS-CRP also checked between two groups

ELIGIBILITY:
Inclusion Criteria:

* all patients who have undergone PCI due to chronic stable angina

Exclusion Criteria:

* Patients with acute coronary syndrome
* Primary LDL>190 mg/DL
* Patients who developed statin-induced myopathy or rhabdomyolysis
* Persistent increase in hepatic enzyme levels or hepatic failure
* Pregnancy and breast feeding
* Statin hypersensitivity
* Patients with history of multiple atherosclerotic events
* Patients who received high intensity statin before the study enrollment.

Ages: 52 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
major adverse cardiovascular events (MACE) | 1 year
  major adverse cardiovascular events
serum level of HS-CRP | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Professor kojuri cardiology clinic, Shiraz, Outside of the US, Iran

IPD SHARING:
Plan to Share IPD: No
Dat available on demand of reviewer